CLINICAL TRIAL: NCT04530201
Title: Developing a Complete Cervical Cancer Screening Solution Based on First-void Urine Self-sampling: Validation for Detection of Precursor Lesions
Brief Title: CASUS: Validation for Detection of Precursor Lesions
Acronym: CASUS-WP4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Novosanis NV (Industry); Self-screen B.V. (Unknown)
Responsible Party: Principal Investigator, Pierre Van Damme, Principal Investigator, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BE3002020000101
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia; Human Papilloma Virus; HPV-Related Cervical Carcinoma; Urine
Keywords: Biomarker; First-void urine; Screening; Triage
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample collection (Other): Women will self-collect two first-void urine samples at home, the day prior to colposcopy. During the colposcopy visit, the clinician will collect an additional cervical smear. Colposcopy and histology results (when available) will be used as reference test.
  Interventions: Device: Colli-Pee Small Volumes (10 mL) device

INTERVENTIONS:
Device: Colli-Pee Small Volumes (10 mL) device — Women will self-collect two first-void urine samples at home the day prior to colposcopy using the new generation Colli-Pee Small Volumes (10 mL) device (Novosanis, Belgium). The collector tube will be prefilled with a non-toxic nucleic acid preservative including an internal process control.

SUMMARY:
The goal of the overall CASUS project is to develop the first fully molecular integrated cervical cancer screening approach, based on first-void urine as an easily accessible and non-invasive source of biomarkers. In contrast to current screening modalities, the CASUS approach will identify women with clinically relevant disease in need of treatment using only a single sample that can be collected at home (one-step triage).

DETAILED DESCRIPTION:
CASUS work package 4 (WP4):

The main aim of this study is to validate the HPV-Risk assay (Self-screen, The Netherlands) followed by multiplex methylation specific quantitative PCR (qMSP, VU University Medical Center, The Netherlands) on first-void urine (Colli-Pee Small Volumes (10 mL) device, Novosanis, Belgium) of HPV positive women for detection of clinically relevant precursor lesions by sampling a cohort of women referred for colposcopy. The number of women in this cohort will allow us to clinically validate the use of the HPV-Risk/qMSP assay in DNA extracts of first-void samples after optimization of sample volume, internal process control, and DNA extraction method (Centre for the Evaluation of Vaccination, University of Antwerp, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Female
* 25 years until 64 years old
* Referred to colposcopy due to a single/multiple (probable) high-risk HPV infection and/or abnormal cervical squamous intraepithelial/glandular lesion.
* Gives informed consent to the research team at the clinical study site to contact his/her general practitioner and/or gynaecologist to access details of the participants HPV test results and cervical screening history.
* Is able to understand the information brochure/what the study is about.

Exclusion Criteria:

* Women that underwent hysterectomy
* Pregnant women
* Treatment for cervical cancer in the last 6 months before participation in the study
* Participating in an interventional clinical study (where e.g. a medical device, drug, or vaccine is evaluated) at the same time of participating in this study. Participation in another observational or low-interventional clinical study at the same time is allowed.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 332 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
HPV DNA (HPV16, HPV18, other high-risk HPV (HPV31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66, -67, and -68)) measured using the HPV-risk assay (Self-Screen BV). | Through study completion, an average of 1 year
  Analytical test results:
  HPV DNA (HPV16, HPV18, other high-risk HPV (HPV31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66, -67, and -68)) concentrations [cycle threshold values] in first-void urine samples from all study participants.
  Clinical test accuracy:
  HPV DNA (HPV16, HPV18, other high-risk HPV (HPV31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66, -67, and -68)) test outcomes [positive, negative] in first-void urine samples from all study participants compared to the gold standard reference test for cervical cancer screening; i.e. histology [Cervical Intraepithelial Neoplasia grade 0-3+].
Methylation ratio of a host cell gene marker panel (PreCursor-U+) measured using quantitative methylation specific PCR (qMSP). | Through study completion, an average of 1 year
  Analytical test results:
  Methylation levels of a host cell gene marker panel (PreCursor-U+) reported in a methylation ratio [(2^-deltaCT *100) with CT being cycle threshold values] in first-void urine samples from all study participants.
  Clinical test accuracy:
  Methylation panel (PreCursor-U+) test outcomes [positive, negative] in first-void urine samples from all study participants compared to the gold standard reference test for cervical cancer screening; i.e. histology [Cervical Intraepithelial Neoplasia grade 0-3+].

SECONDARY OUTCOMES:
Human DNA (GAPDH) | Through study completion, an average of 1 year
  Human DNA (GAPDH) concentrations [cycle threshold values] in first-void urine samples from all study participants measured by quantitative PCR (qPCR).
Internal control DNA (IC DNA) | Through study completion, an average of 1 year
  Internal control DNA (IC DNA) concentrations [cycle threshold values] in first-void urine samples from all study participants measured by quantitative PCR (qPCR).
Human DNA (Beta-globin) | Through study completion, an average of 1 year
  Human DNA (Beta-globin) concentrations [cycle threshold values] in first-void urine samples from all study participants measured using the HPV-risk assay (Self-Screen BV).
Human DNA reference gene (ACTB) | Through study completion, an average of 1 year
  Human DNA reference gene (ACTB) concentrations [cycle threshold values] in first-void urine samples from all study participants measured by quantitative methylation specific PCR (qMSP).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, MD, PhD, Principal Investigator — Universiteit Antwerpen; Alex Vorsters, Ir, PhD, Study Chair — Universiteit Antwerpen; Severien Van Keer, PhD, Study Chair — Universiteit Antwerpen
Locations (3):
- Belgium (3):
  - Vrouwenkliniek - Universitair Ziekenhuis Gent (UZ Gent), Ghent, Oost-Vlaanderen
  - Femicare VZW & Departement Verloskunde & Gynaecologie - Regionaal Heilig Hart Ziekenhuis Tienen, Tienen, Vlaams-Brabant
  - Gynécologie-obstétrique - CHU de Liège, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hendrickx JO, Van Keer S, Donders G, Weyers S, Doyen J, Beyers KCL, Rios-Cortes A, Meers N, Teblick L, Vankerckhoven VVJ. Home-based urinary HPV self-sampling for the detection of cervical cancer precursor lesions: attitudes and preferences from Belgian females participating in the CASUS study. Arch Public Health. 2025 Feb 12;83(1):32. doi: 10.1186/s13690-024-01490-3. PMID 39934916